CLINICAL TRIAL: NCT03391336
Title: Median Nerve Injury in US-guided Carpal Tunnel Injections
Status: Completed | Type: Observational
Sponsor: yi-chih HSU (Other)
Responsible Party: Sponsor-Investigator, yi-chih HSU, Radiologist, Tri-Service General Hospital
Organization: Tri-Service General Hospital (Other)
Other Study IDs: TSGHIRB 2-105-05-110
Record Dates: First submitted 2017-12-23; First posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2017-12

CONDITIONS: Injury of Median Nerve Distal to Forearm; Carpal Tunnel Syndrome
Keywords: Carpal tunnel syndrome; Median nerve injury; Steroids; Ultrasound; Injections
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Carpal tunnel syndrome (CTS) is the most common nerve compression disorder in the upper extremity. It can be treated with surgical or nonsurgical methods. When nonsurgical treatment is indicated, local corticosteroid injection into the carpal tunnel can be used to reduce pain and tingling sensation.

Currently, the most widely used ultrasound (US)-guided CTS-injection method are transverse and longitudinal approach. Although we can accurately place needle within the carpal tunnel using this approach and this approach is easy to learn, median nerve injury (MNI) is still an inevitable complication and difficult to be treat.

MNI is the most serious complication associated with a local corticosteroid injection for CTS among them. A MNI will be presented with shooting pain at the injection time or transient exacerbation of CTS symptoms following the corticosteroid injection because of the pain which often masked by anesthetic during injection. Permanent damage of MN should be considered if the symptoms persist and exacerbate for more than 48 hours. A surgical intervention such as neurolysis, resection or graft repair or a gentle debridement of the crystal from the nerve may be performed in the patients with median nerve damage. Hence, early recognition of MNI before corticosteroid injection may avoid the permanent damage of MN.

Accordingly, the aim of this study is to determine the relationship between the MNI with the possible influencing factors and findings in the US-guided corticosteroid injection for patients with CTS with and to compare the therapeutic efficacy in the patients with and without MNI.

DETAILED DESCRIPTION:
Patients:

This study was approved by our institutional review board (Tri-Service General Hospital); however, patient consent was not required for the retrospective review of records and images because patient anonymity was preserved. The patients with clinically suspected CTS evaluated by the referring neurologist (F. C. Y.), and the clinical tests included (1) typical symptoms, eg, hand numbness and pain in the distribution of the median nerve, nocturnal worsening of symptoms, worsening symptoms while driving or gripping, (2) positive Tinel's and/or Phalen's sign, (3) failure of splinting and/or hand rest. Patients with clinically suspected CTS underwent US examination. The diagnoses of CTS in these patients were confirmed by US and/or electrodiagnostic investigations.

Ultrasonography:

The US was provided using a scanner (Xario 100; Toshiba, Tokyo, Japan) with a 7~18 MHz linear transducer (PLU-1204BT). The US examinations were performed by an experienced technician (C.Y. H.) with 6 years of musculoskeletal experience in US. The technician received specialized training on the procedure used to scan the MN regarding the CTS and to record the images and was directly supervised by the attending radiologist (Y.C.H.). The US images after the US-guided hydrodissection were recorded by the attending radiologist (Y.C.H.). The diagnosis of CTS was based on qualitative US criteria, with a cutoff value of ≥12 mm2 regarding the cross-sectional area (CSA) of the MN (CSA-MN) at the inlet of the carpal tunnel. The diagnoses of CTS were confirmed by electrodiagnostic investigations in the patients with US findings of the CSA-MN < 12 mm2 at the inlet of the carpal tunnel. The flowchart illustrating patient selection is shown in Fig. 1. All US images and the measurements of cross sectional area (CSA) of the median nerve at the inlet of carpal tunnel were saved in the picture archiving and communication system (PACS). All the patients with clinically suspected CTS during the study period were examined using a standardized US protocol previously described to assess the MN at the wrist level (Figure. 1). Within 1 month after US-guided corticosteroid injection, we assessed the MN again with this manner.

Ultrasound needle guidance:

The US-guided injection procedure was performed in a standardized manner. The one-needle two-syringe technique with US guidance was used where (1) one needle is used for anesthesia, hydrodissection, and intra-carpal tunnel injection; (2) the first syringe is used to anesthetize, hydrodissect, and dilate the intra-carpal tunnel space; and (3) the second syringe is used to inject the corticosteroid therapy into the new hydrodissected space (Figure 2). After hydrodissection, the empty lidocaine syringe was detached from the needle while still in the carpal tunnel, and a 3-ml syringe prefilled with 10 mg triamcinolone acetonide suspension was attached to the indwelling needle, and the treatment was slowly injected into the hydrodissected neutral space that was closest to the MN. The injections were performed in a standardized fashion by a musculoskeletal radiologist (Y.C.H.) with 13 years of experience in US.

Smith et al have recommended the needle should be passed above and below the median nerve to fill the injectate around the median nerve with an ulnar approach. Although we can accurately place needle within the carpal tunnel using this ulnar approach and this approach is easy to learn, neurovascular injury may happened in the conditions of well-described anatomic variation (eg, persistent median artery, bifida of MN), and unable supination of wrists. In these patients with difficulty in performing hydrodissection, The investigators may abandon needle redirection deep to the median nerve or chose the radial approach when clearly identifying the fascial passage of the palmar cutaneous branch (PCB) of the MN (Figure 3). The only mater in the radial approach the investigators need attention is the avoidance of damage of the PCB of the MN.

Data collection The patients' medical records were reviewed by a neurologist (F.C.Y.). Routinely, the investigators recorded clinical data (including sex, age, and side of injection, height and weight [which were used to estimate BMI]), complications, and the effect of treatment. Blood in the needle after US-guided hydrodissection was recorded as vascular injury in the US-guided corticosteroid injection. The US images were analyzed by two musculoskeletal radiologists (Y.C.H.) and (G.S.H.) who were blinded to the occurrence of MNI. The investigators determined the absence of hyperechoic rim of MN on pre-injection US, the inter-scan change of nerve echogenicity of MN at the inlet of carpal tunnel in consensus. The investigators determined the swelling of MN including the flattening ratio (largest diameter/smallest diameter) and cross-sectional area at the inlet of carpal tunnel at the time of before and after the hydrodissection on the procedure US. The rater (Y.C.H.) performed duplicate measurements, with the second measurement obtained 2 weeks after the first. All measurements were performed with the aid of a PACS, a mouse pointer (cursor), and automated computer calculation. The mean of two measurements was considered to be the final value.

The investigators hypothesized that multiple pre-injection factors, including sex, age, side of injection, patient BMI, diabetes mellitus, anatomic variation of MN (eg, persistent median artery, bifida of MN), site of needle passed into the skin; and findings after hydrodissection such as vascular injury and the US findings of MN after hydrodissection may have relevance to MNI (Figure 4). To evaluate the relevance of these pre-injection factors to MNI, we decided to convert these continuous variables into dichotomous variables. Subjects were divided into old and young groups on the basis of a cutoff age of 40 years, thin and obese groups on the basis of a cutoff BMI of 30, ulnar and radial approaches groups on the basis of site of needle passed into the skin, hydrodissection in the superficial and deep to the median nerve groups on the basis of needle redirection.

Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) is the most commonly used questionnaire for the measurement of the severity of symptoms and functional status with reproducibility, internal consistency, and validity in patients with CTS. The symptom severity subscale of BCTQ (BCTQs) consists of 11 questions with scores from 1 point (mildest) to 5 points (most severe), and the functional status of BCTQ (BCTQf) subscale is made up of 8 questions with scores from 1 point (no difficulty in activity) to 5 points (unable to perform the activity at all). Patients were seen in the subsequent clinical visit to determine outcomes. The investigators also recorded the decrease of BCTQ between the before and after US-guided corticosteroid injection as decrement of BCTQ.

Statistical analysis All the measurements regarding the change of MN were presented as mean ± standard deviation. Intra-rater agreement was evaluated using the intra-class correlation coefficient (ICC). Fisher's exact test was used to determine the association between MNI to these independent factors before injection and findings after hydrodissection. Receiver operating characteristic (ROC) analysis was used to determine the "cut-off point" for predicting the presence of MNI. The patients with and without the diagnosis of MNI were defined as 2 groups. The therapeutic efficacy of these 2 groups were compared by using a Student t test (for BCTQ before corticosteroid injection, BCTQ after corticosteroid injection, and decrement of BCTQ), as appropriate.

All the statistical tests were performed with the SPSS software (v. 16; SPSS, Inc. Chicago, IL, USA). Significance testing was conducted using a two-tailed alternative hypothesis. Differences were considered statistically significant for a p value of < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* The clinical tests included (1) typical symptoms, eg, hand numbness and pain in the distribution of the median nerve, nocturnal worsening of symptoms, worsening symptoms while driving or gripping, (2) positive Tinel's and/or Phalen's sign, (3) failure of splinting and/or hand rest.
* Patients with clinically suspected CTS underwent US examination.
* The diagnoses of CTS in these patients were confirmed by US and/or electrodiagnostic investigations.

Exclusion Criteria:

* prior carpal tunnel release
* loss of follow-up US examinations
* previous US-guided carpal tunnel injections
* US-guided carpal tunnel injections with recurrence on ipsilateral hands

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with carpal tunnel syndrome in a single center (TSGH)
Sampling Method: Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
The observation of median nerve injury | July 2017 to September 2017
  The investigators observed if patient had symptoms of shooting pain after the corticosteroid injection along with numbness, paresthesia and other sensory deficits and distributions in the median nerve supply area.

SECONDARY OUTCOMES:
The intra-rater agreement of measurements | July 2017 to September 2017
  The investigators determined the intra-rater agreement for these quantitative measurements (flattening ratio and cross-sectional area of the MN) for the before and after hydrodissection US.
The relationship between pre-injection factors and MNI | July 2017 to September 2017
  The investigators determined the associations between MNI and the pre-injection factors. The factors includes sex, age, side of injection, site of needle passed into the skin, BMI, anatomic variation of MN, absence of hyperechoic rim of MN, and whether or not they have diabetes mellitus.
The relationship between post-injection factors and MNI | July 2017 to September 2017
  The investigators determined the associations between MNI and the post-injection factors. The hydrodissection findings includes vascular injury during hydrodissection, altered echogenicity, decrease flattening ratio, and increase cross-sectional area (CSA) of MN on US after hydrodissection.
The symptoms relief after corticosteroid injection in the groups of MNI or not | July 2017 to September 2017
  The investigators observed the symptoms relief, which was rated using a Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) scores.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Chih Hsu, MD, Principal Investigator — IRB of TSGH, Taipei, Taiwan
Locations (1):
- No. 325, Sec. 2, Cheng-kung Rd., Neihu 114, Taipei, Taiwan, R.o.c., Taiwan